CLINICAL TRIAL: NCT01682109
Title: Palatability Testing of a New Paediatric Formulation of Valacyclovir for the Prophylaxis and Treatment of VZV and HSV Infections in Children
Brief Title: Palatability Testing of a New Paediatric Formulation of Valacyclovir
Acronym: VALID-0
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UMCN-AKF 11.05
Record Dates: First submitted 2012-09-05; First posted 2012-09-10 (Estimated); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Varicella Zoster Virus Infection; Herpes Simplex Virus Infection
Keywords: prophylaxis; herpes zoster; herpes simplex; valacyclovir; palatability; paediatric
MeSH Terms: conditions — Varicella Zoster Virus Infection; Herpes Simplex; Herpes Zoster | interventions — Valacyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- new paediatric valacyclovir formulation (Experimental): Newly developed formulation
  Interventions: Drug: Valacyclovir
- reference valacyclovir formulation (Active Comparator): Formulation derived from FDA label information
  Interventions: Drug: Valacyclovir

INTERVENTIONS:
Drug: Valacyclovir
  Other Names: valacyclovir solution

SUMMARY:
Palatability testing of a new paediatric formulation of valacyclovir in children 4-12 years of age and at least one of their parents. Children will be included, who received (val)acyclovir prophylaxis in the past, or will probably need it in the future i.e. children with primary immune deficiency or cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 4 years of age.
* Subject weighs at least 15kg.
* Subject is capable of performing the taste assessment, according to the investigator's judgement.
* The child and parent(s) are willing to participate in the taste assessment.
* Signed informed consent by the legal guardian for participation of the child and if the parent also wants to participate: signed informed consent for their own participation, prior to start of the study.

Exclusion Criteria:

* Documented history of sensitivity/idiosyncrasy to medicinal products or excipients.
* Presence of any condition that influences taste sensation (such as upper respiratory infection, febrile illness within 3 days before the first dose, mucositis or use of medication that influences taste perception, as described in the label information).

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Selection of oral solution with best taste | Day 1
  Patients (children) will assess the taste of 3 different oral solutions. A questionnaire has to be completed to order the palatability of the three formulations.

SECONDARY OUTCOMES:
Taste assessment | Day 1
  Children will score the taste of 3 different oral valacyclovir solutions. A 100 mm facial hedonic scale will be employed to indicate the palatability of each formulation.
Predictability of palatability preference of the child by parents. | Day 1
  To determine whether parents can predict the palatability preference of their child.

CONTACTS AND LOCATIONS:
Overall Officials: David Burger, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Center, Nijmegen, Netherlands

REFERENCES:
- [Result] Bastiaans DET, Immohr LI, Zeinstra GG, Strik-Albers R, Pein-Hackelbusch M, van der Flier M, de Haan AFJ, Boelens JJ, Lankester AC, Burger DM, Warris A. In vivo and in vitro palatability testing of a new paediatric formulation of valaciclovir. Br J Clin Pharmacol. 2017 Dec;83(12):2789-2797. doi: 10.1111/bcp.13396. Epub 2017 Sep 20. PMID 28800385